CLINICAL TRIAL: NCT05386836
Title: Single-center Study Assessing the SpO2 and Pulse Rate Accuracy of the Sunrise Sensor 2 Compared to Arterial Blood Samples Oxygen Saturation Assessed by CO-oximetry and ECG Respectively, Under Non-motion Conditions in Healthy Adults
Brief Title: The Sunrise SpO2 and Pulse Rate Accuracy Validation Study
Acronym: S2-SOPRAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunrise (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-367
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Validation Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adult volunteers (Experimental): All subjects within this single arm of the study will undergo the validation experiment as described in the description
  Interventions: Device: Pulse oximeter validation population

INTERVENTIONS:
Device: Pulse oximeter validation population — Evaluation of the SpO2 accuracy performance of the Sunrise Sensor 2 placed at the tip of the chin during non-motion conditions over the range of 70-100% by comparison to SaO2 values determined from arterial blood sample specimen analyzed by a CO-oximeter.

SUMMARY:
The purpose of this study is to evaluate the SpO2 accuracy performance of the Sunrise Sensor 2 placed at the tip of the chin during non-motion conditions over the range of 70-100% by comparison to SaO2 values determined from arterial blood sample specimen analyzed by a CO-oximeter. Testing is conducted under normal office environment conditions. It is expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system will meet the required specification of ARMS of 3.5% or less allowed for reflectance technology in non-motion conditions for the range of 70-100% SaO2.

A secondary goal is to evaluate the pulse rate performance simultaneously collected over the SpO2 range covered.

DETAILED DESCRIPTION:
Subjects will be given medical grade mixtures of oxygen and nitrogen to induce stable plateaus across the range of 100% to 70% SaO2. When the reference system's blood saturation stabilizes at an acceptable plateau level, blood sampling can start. Four to eight arterial blood samples will be collected for each plateau, while keeping at least 20 seconds in between each sample and at least 30 seconds once the plateau has been reached. The blood will be immediately analyzed by the reference CO-Oximeter to measure the arterial oxygen saturation (Functional SaO2). SpO2 values from the Sunrise sensor 2 will be collected electronically simultaneously to blood drawn from the indwelling catheter. Data will be collected under non-motion conditions. The pulse rate will be simultaneously collected over the SpO2 range covered. The reference method for the computation of pulse rate accuracy will be an ECG heart rate. The total duration of the test will be about 1 hour per subject. Data analysis results will provide documentation showing SpO2 and pulse rate accuracy performance of the Sunrise sensor 2 as compared to arterial blood samples measured by Reference CO-Oximetry and to ECG heart rate, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with positive Allen's test
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study
* 15% of the study population or 2 subjects (whichever is larger) with dark pigmented skin should be included in the study

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study
* Subjects with known heart or cardiovascular conditions
* Subjects with other known health condition (diabetes, thyroid disease, kidney disease/chronic renal impairment, history of seizures (except childhood febrile seizures) or epilepsy, or unexplained syncope, recent history of frequent migraine headaches, recent head injury, cancer/chemotherapy)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
SpO2 ARMS determination | Within 1 month after subject recruitment
  SpO2 accuracy root-mean-square (ARMS) determination for the range of 70- 100%., i.e., the RMS difference between measured values and reference values.

SECONDARY OUTCOMES:
Pulse rate ARMS determination | Within 1 month after subject recruitment
  Pulse rate accuracy root-mean-square (ARMS) determination

CONTACTS AND LOCATIONS:
Locations (1):
- Respisom, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No